CLINICAL TRIAL: NCT06785792
Title: Validity and Reliability of Artificial Intelligence-Assisted Posture Applicatıon in Young Adults
Brief Title: Artificial Intelligence-Assisted Posture Applicatıon
Status: Recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Prof.Dr, Izmir Democracy University
Other Study IDs: Izmir Democracy
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Postural; Defect
Keywords: posture; validity; reliability; artificial intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: The population of the research consists of young adult individuals in the general Turkish population, and the research sample consists of young adult individuals in the Turkish population who volunteered to participate in the research. There is only one research group consisting of volunteer individuals.

SUMMARY:
Posture is defined as the situation in which each part of the body is properly positioned in the adjacent segment and is in the most ideal position in proportion to the whole body. Posture requires the appropriateness of joint combinations and positions during movement. With the development of technology, various phone and computer-aided applications are used both in the correction and evaluation of posture. It is thought that posture disorders may cause various pathological problems in the future and may lead to functional limitations in the individual. With the developing technology, there are a limited number of studies on the validity and reliability of phone and computer-aided applications in every field of health. The aim of this study is to perform the validity and reliability study of a sensorless objective application integrated with artificial intelligence used in posture evaluation with the developing technology.

DETAILED DESCRIPTION:
Posture is defined as the situation in which each part of the body is properly positioned in the adjacent segment and is in the most ideal position in proportion to the whole body. Posture requires the appropriateness of joint combinations and positions during movement. Genetics, the environment in which the individual lives, physical condition, socio-economic level, emotional state, and physiological changes that the individual undergoes during the growth and development process are important intrinsic and extrinsic factors that determine posture. The main purpose of posture analysis is to identify the patient's current postural deviations and to develop appropriate treatment programs and also to evaluate possible changes. In posture analysis, tools such as pendulums, special pens for marking vertebrae, tape measures, rulers, posture boards or wooden blocks are used. When performing posture analysis, the person should be wearing appropriate clothing and their feet should be bare; the analysis is performed when the person is in the position they feel most comfortable in. Posture analysis is performed from three different directions: from the front (anterior), from the side (lateral), and from the back (posterior). There are different methods for posture analysis. These methods can be interpreted with numerical and verbal data. There are also methods where not only the whole body but also body segments can be evaluated separately. In posture analysis, observational methods, New York State and Bragg posture table and head-neck and shoulder girdle, sagittal plane photography method, symmetrygraph, lateral radiography, distance measurements, goniometric measurements are some of these methods. In a study conducted to determine the relationship between posture, pain, upper extremity functions, and anxiety levels with various parameters in musicians, the Posture Screen Mobile (PSM) application with an ICC score of 0.71-0.99 was used, while in another study investigating the effect of posture on health-related quality of life in young adults, the Reedco Posture Score with an ICC score of 0.85-0.95 was used. It is seen that New York Posture Analysis is used in studies evaluating the posture of school-age children and young adults. In a study evaluating the effect of posture correction applications on neck pain and function on smartphones, it is seen that there are applications on phones for posture correction applications. This situation shows us that with the development of technology, various phone and computer-supported applications are also used in both posture correction and evaluation. It is thought that posture disorders can cause various pathological problems in the future and cause functional limitations in the individual. With the developing technology, there are a limited number of studies on the validity and reliability of phone and computer-supported applications in every field of health. The aim of this study is to carry out the validity and reliability study of a sensorless objective application integrated with artificial intelligence used in posture evaluation with the developing technology.

ELIGIBILITY:
Inclusion Criteria:

* Young adult individuals between the ages of 18-39
* Individuals who volunteer to participate in the study
* Individuals who are Turkish citizens, reside in Turkey and have been in Turkey for at least 1 month before and during the study period
* Individuals who can communicate in written and verbal Turkish

Exclusion Criteria:

* Individuals with any physical or mental disability and/or cognitive impairment
* Pregnant women
* Individuals with orthopedic, neurological, vestibular diseases that may affect walking and balance functions
* Individuals with neuromuscular system diseases or diseases that will prevent postural control measurements (vertigo, neuropathy, etc.) or those using medication

Ages: 18 Years to 39 Years | Sex: All
Age Groups: Adult
Study Population: The population of the research consists of young adult individuals in the general Turkish population, and the research sample consists of young adult individuals in the Turkish population who volunteered to participate in the research. There is only one research group consisting of volunteer individuals. There is only one research group within the scope of the study.
  Data will be collected from individuals face to face. Individuals who meet the inclusion criteria and volunteer will be evaluated simultaneously by 3 expert physiotherapists on consecutive days (3 days) at the same time, with 3 repetitions using observational posture analysis, New York posture scale and artificial intelligence-supported posture application.
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Posture Evaluation System (Fizyosoft™ Becure Posture System) | Individuals who meet theinclusion criteria and volunteer will be evaluated simultaneously by 3 expert physiotherapists on consecutive days (3 days) at the same time, with 3 repetitions using Posture Evaluation System (Fizyosoft™ Becure Posture System).
  Becure Posture is an artificial intelligence-supported technological solution that allows individuals to perform posture analysis, can be used via mobile devices or computer applications. The purpose of the application is to perform posture analysis by adding photographs of clients or patients, to provide analysis by physically taking their photographs, to automatically determine joint points with artificial intelligence support and to enable users to manually edit these points when needed. It also allows users to receive reports. The application is licensed and can be accessed from AppleStore or PlayStore after obtaining the license. After logging in to the account, a total of 4 photos must be uploaded to the page that opens, including the name and surname, in order to evaluate the posture: anterior, posterior, right lateral and left lateral. After the photo is uploaded, a report is printed out in which the detailed posture analysis of the upper and lower extremities is performed.

SECONDARY OUTCOMES:
New York Posture Assessment | Individuals who meet theinclusion criteria and volunteer will be evaluated simultaneously by 3 expert physiotherapists on consecutive days (3 days) at the same time, with 3 repetitions using New York Posture Assessment.
  NYPD evaluates the correct and incorrect alignment of various body parts of a person in an anatomical position using a quantitative approach. A scoring system is used in the assessment. In the posture scoring, 5 points are given if it is correct, 3 points if there is a moderate disorder and 1 point if there is a high degree of disorder. The total score obtained as a result of the scoring is a maximum of 65 and a minimum of 13. In the developed standard evaluation criteria, if the total score is ≥45, it is defined as very good, 40-44 as good, 30-39 as medium, 20-29 as weak, and ≤19 as bad. A high score indicates that the posture is correct.
Posture Analysis with Static Observation (Lateral, Anterior, Posterior) | Individuals who meet the inclusion criteria and volunteer will be evaluated simultaneously by 3 expert physiotherapists on consecutive days (3 days) at the same time, with 3 repetitions using observational posture analysis
  Posture analysis performed with static observation is performed in 3 aspects: lateral posture analysis, anterior posture analysis and posterior posture analysis. Observed disorders will be recorded by scoring between 0-3. In the scoring system, 0 indicates no, 1 indicates mild, 2 indicates moderate and 3 indicates severe disorders.
Demographic Information Form | baseline
  With this form, information about the age, gender, height, weight, pregnancy status, educational status, occupation, smoking and alcohol use status, bag carrying style that may affect posture, frequency of computer use, study time, sports of interest and the duration of performing the sports of interest will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Prof.Dr, Principal Investigator — İzmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Karabağlar/İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fortin C, Feldman DE, Cheriet F, Labelle H. Clinical methods for quantifying body segment posture: a literature review. Disabil Rehabil. 2011;33(5):367-83. doi: 10.3109/09638288.2010.492066. Epub 2010 Jun 23. PMID 20568973
- [Background] Czakwari A, Czernicki K, Durmala J. Faulty posture and style of life in young adults. Stud Health Technol Inform. 2008;140:107-10. PMID 18810009
- [Background] Szucs KA, Brown EVD. Rater reliability and construct validity of a mobile application for posture analysis. J Phys Ther Sci. 2018 Jan;30(1):31-36. doi: 10.1589/jpts.30.31. Epub 2018 Jan 27. PMID 29410561